CLINICAL TRIAL: NCT06347107
Title: Robotic Subretinal tPA Injection Study
Acronym: RoTIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: DORC Dutch Ophthalmic Research Center International BV (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S67215
Record Dates: First submitted 2024-03-21; First posted 2024-04-04 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Subretinal Hemorrhage; Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Intervention Model Description: Investigator-initiated, academic, mono-center, prospective, interventional case study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Robotic subretinal tPA injection group (Experimental): The purpose of this study is to determine the feasibility of subretinal injection of tPA assisted by a prototype robotic device.
  Interventions: Device: Robotic subretinal tPA injection

INTERVENTIONS:
Device: Robotic subretinal tPA injection — -The insertion of a 41G subretinal needle adjacent to a subretinal hemorrhage using the stabilizing (tremor-reducing) properties of a robotic instrument in order to slowly inject tPA and evaluate whether the needle can be held in place for up tot 3 minutes.

SUMMARY:
In the RoTIS study, the investigators would like to test the robotic stabilizer for the subretinal injection of tPA in patients with subretinal hemorrhage during standard-of-care surgery. The surgical devices used during this procedure will be the following:

* The robotic stabilizer (prototype - FAMHP approval received)
* 41G subretinal needle (CE marked - used within label)
* Inicio micro-injection system (CE marked - used within label) The Inicio system mounted with the 41G needle will be held by the robot, and guided by the surgeon towards the required position. When the tip of the needle is in the desired subretinal position, the robotic stabilizer will be locked and the tPA will be injected till sufficient subretinal bleb formation is obtained, with a maximal duration of up to 3 minutes.

As performed routinely, the surgical view through the microscope will be video-recorded and while the injection is being administered, the built-in iOCT of the Artevo surgical microscope (Zeiss, Oberkochen, Germany) will be used to scan the retina area around the injection site to record the subretinal bleb formation for later review.

DETAILED DESCRIPTION:
Age-related macular degeneration is a common disease in the elderly population. In the atrophic form, central retinal degeneration leads to the formation of central metamorphopsia or scotoma. In 10% of all cases, the atrophic form becomes proliferative, whereby newly formed vessels grow under the macular area. Although this proliferation can be controlled in most patients with intravitreal injections of anti-VEGF, in some cases a subretinal hemorrhage occurs which causes a drastic drop in visual acuity.

Before anti-VEGF treatment existed, removal of the subretinal vessels followed by a macular translocation or transplantation of retinal pigment epithelium cells was sometimes considered in such cases when the second eye became affected 1,2.

Later on, when anti-VEGF and other growth inhibiting products became available (Macugen, Lucentis, Avastin, Eylea, BeoVue), ophthalmologistsdeveloped a far less invasive surgically technique to inject tPA subretinally into the blood clot using a 41G (0.11mm) subretinal needle, followed by an air fill of the vitreous cavity to displace the subretinal liquefied blood away from the macular area 3,4.

Since the causal neovascular vessels are not removed during this procedure, repeat injections with anti-VEGF or analogue products are mandatory afterwards to reduce the risk of recurring hemorrhage.

This surgical technique typically consists of a standard three-port pars plana vitrectomy, induction of posterior vitreous detachment (if not already present), core and peripheral vitrectomy (EVA Nexus surgical system, DORC, Zuidland The Netherlands). Macular detachment is induced by subretinal injection of a balanced salt solution (BSS). The injection device is a 41G polyimide straight subretinal cannula with 27G shaft (DORC) connected to the Inicio micro-injection system (DORC). The EVA Nexus surgical system, the 41G subretinal needle and the Inicio micro-injection system used in this study are all CE-labeled devices and used on-label.

This surgical technique has been previously described in the literature3,4 albeit performed using older generations surgical systems, the Associate and EVA, respectively (DORC, Zuidland, The Netherlands). In our department, such surgical procedure with subretinal injection of tPA is performed about 25 times yearly.

More recently, gene therapy is being developed to treat several different congenital eye diseases. In 2021, the first of such products became commercially available (Luxturna, Novartis). All the gene therapy vehicles which are either already available or are being developed have in common that they need to be precisely subretinally injected in a very small volume. For Luxturna application, the standard-of-care is to manually hold the subretinal needle into the subretinal space and to ask the surgical assistant to manually inject the product under the retina while the surgeon holds still the subretinal needle. It does not need to be explained that such surgical conditions are far from ideal to inject a product that costs Eur 375 000 per dose.

A tool that would help the surgeon to eliminate hand-tremor and to hold still the subretinal needle in the subretinal space would be very much welcomed as adjunct in this type of surgery. There is a robotic system available with the CE-mark for intra-ocular surgery (Preceyes, Eindhoven, The Netherlands, recently acquired by Zeiss, Oberkochen, Germany), but this was developed as an aiding tool for intra-ocular membrane peeling. Other systems are being developed but not yet commercially available (eg. Accusurgical, Montpellier, France or Foresight Robotics, Yokn'am Illit, Israel).

In 2017, after more than 10 years of development, the investigators performed robot-assisted retinal vein cannulation with injection of Ocriplasmin during vitrectomy surgery in 4 patients to treat central retinal vein occlusion (study S58782)5. For that study, a robotic stabilizer was used that has two main functions while holding a surgical instrument:

* It removes high-frequency movements from the surgeons' hand thereby offering a tremor-dampening feature.
* It can be locked when the tip of the instrument (needle) is in the desired position allowing a prolonged injection of liquid (medication) over several minutes while the tip remains in the same position It must be emphasized here that our robotic stabilizer is used as a co-manipulation system: the surgical instrument is held by both the surgeon and the robot, therefore guaranteeing that the surgeon has always has control and override possibility. This in contrast with almost all other robots for eye surgery that are available or under development which are tele-manipulating devices. In such device, the surgeon holds joysticks to remotely control the robot that holds the surgical instrument, similar to the Da Vinci system, the well-known robot for more general surgery.

During that cannulation study, three devices were under investigation (not CE-labeled):

* The robotic stabilizer
* The study drug (Ocriplasmin - Jetrea)
* The (glass) needle to penetrate the occluded retinal vein In all four patients of trial S58782, the investigators were able to successfully introduce the needle into the occluded vessel, and to inject ocriplasmin for up to 9 minutes long while the robotic stabilizer held the needle in the vessel5.

In the RoTIS study, the investigators would like to test the robotic stabilizer for the subretinal injection of tPA in patients with subretinal hemorrhage during standard-of-care surgery. The surgical devices used during this procedure will be the following:

* The robotic stabilizer (prototype - FAMHP approval received)
* 41G subretinal needle (CE marked - used within label)
* Inicio micro-injection system (CE marked - used within label) The Inicio system mounted with the 41G needle will be held by the robot, and guided by the surgeon towards the required position. When the tip of the needle is in the desired subretinal position, the robotic stabilizer will be locked and the tPA will be injected till sufficient subretinal bleb formation is obtained, with a maximal duration of up to 3 minutes.

As performed routinely, the surgical view through the microscope will be video-recorded and while the injection is being administered, the built-in iOCT of the Artevo surgical microscope (Zeiss, Oberkochen, Germany) will be used to scan the retina area around the injection site to record the subretinal bleb formation for later review.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
2. Patients that are scheduled for vitrectomy surgery to treat a submacular hemorrhage with subretinal injection of tPA.
3. Both vitrectomy-only and combined phaco-vitrectomy surgeries
4. General anesthesia

Exclusion Criteria:

1. Patients aged < 18 years
2. Any disorder, which in the investigator's opinion might jeopardise participant's safety or compliance with the study protocol.
3. Vitrectomy surgery for other indication than mentioned above
4. No post-operative week 8 visit is anticipated
5. General anesthesia not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-06-21 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with succesful subretinal insertion of the robot-held 41G needle | During surgery, once vitrectomy is completed, pass/fail event.
  The insertion of a 41G subretinal needle adjacent to a subretinal hemorrhage using the stabilizing (tremor-reducing) properties of a robotic instrument will be evaluated. Succesful formation of a subretinal bleb will prove that the needle was introduced subretinally. This will be monitored visually through the operating microscope and with intra-operative OCT confirming the bleb formation.
Percentage of patients with stable subretinal position of the needle for at least 3 minutes. | During surgery, immediately after insertion of the needle in the subretinal space for up to 3 minutes.
  The ability to hold the needle still in the subretinal space for a time of up to 3 minutes after initiating bleb formation will be determined.This will be monitored visually through the operating microscope and with intra-operative OCT confirming the stable position of the needle.

SECONDARY OUTCOMES:
Device-related adverse events | Duration of surgery: +/- 90 minutes
  Recording the incidence of device-related adverse events
Functional outcome | 2 months post-operative
  Visual acuity will be compared to a historical cohort of patients undergoing subretinal tPA injection without the help of a robotic arm.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stalmans, MD PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No